CLINICAL TRIAL: NCT03706859
Title: Comparison Between Two Mathematical Methods to Estimate Arterial Occlusion Pressure and Tourniquet Effectiveness in Lower Limb Surgery: Randomized Comparative Study
Brief Title: Two Mathematical Methods to Estimate Arterial Occlusion Pressure and Tourniquet Effectiveness in Lower Limb Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa A. Kasem, Associate professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FM-BSU REC 005/2018
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet inflation pressure method 1 (Experimental): the pneumatic tourniquet inflation pressure at 20 mmHg above the arterial occlusion pressure which will be estimated using the equation of Unver B. et al.,: (AOP=[SBP+10]/KTP)
  Interventions: Procedure: Pneumatic tourniquet inflation pressure
- Tourniquet inflation pressure method 2 (Active Comparator): the pneumatic tourniquet inflateion pressure at 20 mmHg above the arterial occlusion pressure which will be estimated using the equation of Hong-yun Liu et al.,: (AOP = 17.986 + 3.158X1 + 0.408X2)
  Interventions: Procedure: Pneumatic tourniquet inflation pressure

INTERVENTIONS:
Procedure: Pneumatic tourniquet inflation pressure — Pneumatic tourniquet inflation pressure estimation using two different mathematical equations

SUMMARY:
Pneumatic tourniquets are widely used not only to reduce blood loss and to ensure optimal operating conditions during extremity surgery, but also in regional anesthesia (local intravenous) vein puncture and to control life or limb threatening conditions. However, compression of the tissues under a tourniquet is associated with soft tissue damage involving the skin, vessels, muscles, and most importantly, nerves, and are commonly pressure related and can be affected by tourniquet time as well. Therefore, the "minimal tourniquet inflation pressure" necessary to provide a bloodless field has been suggested to minimize the risk of complications from excessive inflation pressure. Arterial occlusion pressure (AOP) is the lowest pneumatic tourniquet inflation pressure required to stop the arterial blood flow into the limb, and its usage has been shown to be useful in optimizing tourniquet cuff pressures. The pressure to which a pneumatic tourniquet cuff should be inflated depends on a number of variables, including the patient's age, skin, blood pressure and the shape and size of the extremity in question, as well as the dimensions of the cuff. One of the estimation method for AOP is based on systolic blood pressure (SBP) and tissue padding coefficient (KTP) values (AOP=[SBP+10]/KTP) according to extremity circumferences. Unver B. et al., used this method to estimate effective tourniquet pressure in total knee replacement under hypotensive general anesthesia tourniquet pressure achieved was 169.7±7.9 mmHg, while Tuncali et al., tested it again in different lower limb surgeries under general or neuraxial anesthesia with normotensive techniques and the achieved maximal tourniquet pressures used was 173.3±15.6 mmHg. Hong-yun Liu et al., established a new occlusion pressure mathematical model for the upper limb based on the correlation analysis between several possible influencing parameters and the minimal pneumatic tourniquet pressure.

DETAILED DESCRIPTION:
After ethical committee approval and informed consent from the patients, 80 adult patients 18-40 years old, (ASA I-II), scheduled for knee arthroscopy under general anesthesia with pneumatic tourniquet around the thigh, will be randomly allocated (using closed opaque envelop) into one of two groups:

* Group (A): where the pneumatic tourniquet inflated 20 mmHg above the arterial occlusion pressure which will be estimated using the equation of Unver B. et al., [1]: (AOP=[SBP+10]/KTP)
* Group (B): where the pneumatic tourniquet inflated 20 mmHg above the arterial occlusion pressure which will be estimated using the equation of Hong-yun Liu et al., [2]: (AOP = 17.986 + 3.158X1 + 0.408X2) Patients will be excluded from the study if they are outside the age range, hypertensive, diabetic, complaining of any lower limb claudications, any vascular disease, hemolytic blood disorders or hypercoagulability.

Upon arrival to the operating room, standard monitoring will be attached (5 lead ECG, pulse oximeter and non-invasive blood pressure) followed by a wide-bore canula will be inserted a big vein in the upper limb. General anesthesia will be induced using fentanyl 1 mcg/kg and propofol 2-3 mg/kg laryngeal mask airway device will be inserted after atracurium 0.5 mg/kg and lungs will be mechanically ventilated to maintain end-tidal CO2 at 36-40 mmHg and maintenance of anesthesia will be achieved using isoflurane 1-2 volume %. Hemodynamic stabilization will be assured and systolic blood pressure will be maintained within the pre-induction values ± 20% using intravenous fluid infusion and titration of inhalational anesthetics.

In all patients, the thigh circumference will be measured 20 cm proximal to the superior pole of the patella then, pneumatic the tourniquet cuff will be placed (deflated) around the thigh with the distal edge 15 cm proximal to the proximal pole of the patella. The tissue padding coefficients based on limb circumferences will be calculated in all patients of group (A) according to table (1) [3].

After three successive stable systolic blood pressure reading (5 minutes apart), an initial systolic blood pressure [initial SBP] reading will take and estimated arterial occlusion pressure (AOP) will be quickly calculated according to one of the previously mentioned equation followed limb exsanguination using an Esmarch bandage, then the tourniquet cuff will be inflated to a safety margin pressure 20 mmHg above the calculated (AOP) [3] which will be the [initial tourniquet pressure]. The time between the initial SBP taking and tourniquet inflation will be measured [initial SBP-to- tourniquet inflation time]. The absence of arterial flow in the lower limb is assured using Doppler probe (HD, Philips) positioned, by an independent anesthetist, at either the dorsalis pedis artery or the posterior tibial artery on the foot to monitor arterial flow distal to the tourniquet. If any arterial flow sound will be heard, the estimated tourniquet pressure will be considered insufficient and the patient will excluded from the study. When no arterial blood flow is secured, the surgeon (blinded to the groups) will allowed to start and will be asked to rate the bloodless surgical field using a 4-point scale [1 (Excellent) = No blood in the surgical field, 2 (Good) = Some blood in the surgical field but no interference with surgery, 3 (Fair) = Blood in the surgical field but no significant interference with surgery, 4 (Poor) = Blood in the surgical field obscures the view] [3] at the beginning, in the middle, and at the end of the surgical procedure.

During the surgery, systolic blood pressure will be measured every 5 minutes and the tourniquet inflation pressure will be always kept 20 mmHg above the SBP.

Surgical procedure and anesthetic management were performed by the same surgical and anesthesia teams respectively. The attending anesthesiologist was aware of the allocated group, but the data analyst, surgeon and the patients were blinded to group allocation.

All the patients will be examined one day after surgery for any complications associated with the tourniquet, (e.g. tissue damage, nerve palsy, lower limb blood flow).

The following will be measured:

* Patient's age, weight and gender and lower limb circumference?
* Operative duration and tourniquet time.
* Initial SBP-to- tourniquet inflation time
* Primary outcome: initial and maximal SBP, initial and maximum tourniquet inflation pressure.
* Secondary outcome: surgeon rating of the bloodlessness of the surgical field.
* Any tourniquet associated complications.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-40 years old, (ASA I-II), scheduled for knee arthroscopy under general anesthesia with pneumatic tourniquet around the thigh,

Exclusion Criteria:

* outside the age range, hypertensive, diabetic, complaining of any lower limb claudications, any vascular disease, hemolytic blood disorders or hypercoagulabilty.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure, | baseline and maximum inflation
  initial and maximal Systolic Blood Pressure,
tourniquet inflation pressure. | baseline and maximum inflation
  initial and maximum tourniquet inflation pressure.

SECONDARY OUTCOMES:
surgeon rating of the bloodlessness of the surgical field. | middle and end of surgery
  surgeon rating of the bloodlessness of the surgical field.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University, Faculty of medicine, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Unver B, Karatosun V, Tuncali B. Effects of tourniquet pressure on rehabilitation outcomes in patients undergoing total knee arthroplasty. Orthop Nurs. 2013 Jul-Aug;32(4):217-22. doi: 10.1097/NOR.0b013e31829aef2a. PMID 23881019
- [Background] Liu HY, Guo JY, Zhang ZB, Li KY, Wang WD. Development of adaptive pneumatic tourniquet systems based on minimal inflation pressure for upper limb surgeries. Biomed Eng Online. 2013 Sep 23;12:92. doi: 10.1186/1475-925X-12-92. PMID 24053348
- [Background] Tuncali B, Boya H, Kayhan Z, Arac S, Camurdan MA. Clinical utilization of arterial occlusion pressure estimation method in lower limb surgery: effectiveness of tourniquet pressures. Acta Orthop Traumatol Turc. 2016;50(2):171-7. doi: 10.3944/AOTT.2015.15.0175. PMID 26969952
- [Derived] Kasem SA, Al Menesy T, Badawy AA, Abd Elmawgoud A, Adel G, Badawy YA. Comparison between two mathematical methods to estimate arterial occlusion pressure and tourniquet effectiveness in lower limb surgery: a prospective, randomized, double blind, comparative study. J Clin Monit Comput. 2020 Aug;34(4):675-681. doi: 10.1007/s10877-019-00366-0. Epub 2019 Jul 25. PMID 31346900